CLINICAL TRIAL: NCT06450145
Title: A Study to Explore the Efficacy and Safety of Interferon-α Combined With ATO and Venetoclax in the Treatment of Arsenic-resistant Acute Promyelocytic Leukemia
Brief Title: Evaluate the Efficacy and Safety of Interferon-α Combined With ATO in the Treatment of Arsenic-resistant APL
Acronym: APL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YJKY20230026
Record Dates: First submitted 2024-04-30; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Tumour
Keywords: APL; arsenic-resistant relapse; interferon α-2b
MeSH Terms: conditions — Neoplasms | interventions — Introns; Arsenic Trioxide; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interferon α-2b (Experimental): Eligible APL patients with arsenic-resistant relapse will enter the run-in period, and the subjects in the run-in phase will be treated with arsenic combined with venetoclax. After the run-in period, the patients were treated with interferon α-2b, arsenic trioxide for injection and venetoclax
  Interventions: Drug: interferon α-2b

INTERVENTIONS:
Drug: interferon α-2b — Eligible APL patients with arsenic-resistant relapse will enter the run-in period, and the subjects in the run-in phase will be treated with arsenic combined with venetoclax. After the run-in period, the patients were treated with interferon α-2b, arsenic trioxide for injection and venetoclax until the outcome of CR/PR/PD/ death/withdrawal/loss to follow-up occurred. Tumor assessments were performed every 4 to 6 weeks (as determined by the investigator) during trial treatment. Those who achieved CR/PR/PD/ withdrawal were then returned to standard treatment (treatment regimen was determined by the clinician), and those who completed the combination treatment period of the trial entered the survival follow-up period.
  Other Names: arsenic trioxide; venetoclax

SUMMARY:
This study was a single-arm, open study. After the screening period, arsenic-resistant APL patients were treated with interferon α-2b, arsenic and venetoclax. The efficacy (ORR) and safety were evaluated.

DETAILED DESCRIPTION:
Eligible APL patients with arsenic-resistant relapse will enter the run-in period, and the subjects in the run-in phase will be treated with arsenic combined with venetoclax. After the run-in period, the patients were treated with interferon α-2b, arsenic trioxide for injection and venetoclax until the outcome of CR/PR/PD/ death/withdrawal/loss to follow-up occurred. Tumor assessments were performed every 4 to 6 weeks (as determined by the investigator) during trial treatment. Those who achieved CR/PR/PD/ withdrawal were then returned to standard treatment (treatment regimen was determined by the clinician), and those who completed the combination treatment period of the trial entered the survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.
* 2. Age 18-70 years old (including boundary value);
* 3. The presence of promyelocytic leukemia-retinoic acid receptor alpha (PML-RARα) confirmed by morphological features, cytogenetic analysis, and real-time quantitative polymerase chain reaction (qPCR);
* 4. Arsenic relapse resistant patients: patients who had relapsed (including molecular relapse) after remission with ATO in the previous treatment, and could not be relieved after standard treatment;
* 5. Eastern Cooperative Oncology Group (ECOG) performance status score 0-2;
* 6. The expected survival time is more than 3 months.

Exclusion Criteria:

* 1. Allergy or contraindication to any study drug involved in the protocol;
* 2. Physical examination, electrocardiogram, laboratory examination, vital signs and test related abnormalities are clinically significant (subject to clinician's judgment);
* 3. Other serious conditions that may limit the patient's participation in the trial, such as severe liver or kidney disease; "Patients with advanced infection, uncontrolled diabetes mellitus, severe cardiac dysfunction (e.g., clinically significant prolongation of the QT interval, potentially fatal torsades de pointes) or a history of angina or major heart disease, autoimmune diseases (as judged by the clinician);"
* 4. Pregnant or lactating women;
* 5. Epilepsy and central nervous system dysfunction;
* 6. Active hepatitis B, active hepatitis A, HIV positive;
* 7. Participate in other clinical trials at the same time
* 8. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 4 to 6 weeks
  Efficacy: objective remission rate

SECONDARY OUTCOMES:
Adverse Events | Through study completion, an average of 1 year
  Safety: the incidence and severity of adverse events were evaluated according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 5.0).
DFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  disease free survival
OS | From date of randomization until the date of date of death from any cause, assessed up to 5 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ping Huang, Study Chair — Zhejiang Provincial People's Hospital; Xiaogang Wang, Study Chair — Zhejiang Provincial People's Hospital
Locations (2):
- China (2):
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No